CLINICAL TRIAL: NCT02698072
Title: Improvement in Pain and Function Following a Therapeutic Exercise Program and Dry Needling in Older Adults With Knee Osteoarthritis: A Randomized Double-blind Multicenter Controlled Clinical Trial
Brief Title: Improvement in Pain and Function Following a Physiotherapy Program in Older Adults With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Ilustre Colegio Profesional de Fisioterapeutas de la Comunidad de Madrid (Unknown)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13/2015
Record Dates: First submitted 2016-01-04; First posted 2016-03-03 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Knee Osteoarthritis
Keywords: Stiffness; Pain; Disfunction
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Exercise Therapy; Dry Needling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise and dry needling (Experimental): 24 therapeutic exercise sessions (twice a week) of a land-based therapeutic exercise program consisting of aerobic exercise (20-25 min warm-up), lower limbs muscle strengthening (20-25 min) and lower limbs muscles stretching (10-15 min).
  6 dry needling sessions (once a week) at all the pain points of the involved symptomatic lower limb/s using Hong's fast-in and fast-out technique with multiple rapid needle insertion.
  Interventions: Other: Therapeutic exercise; Device: Dry needling
- Exercise and sham dry needling (Active Comparator): 24 therapeutic exercise sessions (twice a week) of a land-based therapeutic exercise program consisting of aerobic exercise (20-25 min warm-up), lower limbs muscle strengthening (20-25 min) and lower limbs muscles stretching (10-15 min).
  6 sham dry needling sessions (once a week) at all the pain points of the involved symptomatic lower limb/s using a park sham device consists of a base with a hole in the centre and sticky tape on the bottom. From the top of the base extends a double tube, continuing the central hole in the base.
  Interventions: Other: Therapeutic exercise; Device: Sham dry needling

INTERVENTIONS:
Other: Therapeutic exercise — 20-25 minutes aerobic exercise, 20-25 minutes strength exercise and 10-15 minutes stretch exercise.
Device: Dry needling — Dry needling needle AGUPUNT®
  Arms: Exercise and dry needling
Device: Sham dry needling — Sham dry needling DONGBANG-ACUPRIME®
  Arms: Exercise and sham dry needling

SUMMARY:
This study evaluates the combination of a therapeutic exercise program and dry needling in the treatment of knee osteoarthritis in older adults. Half of participants will receive therapeutic exercise program and dry needling in combination, while the other half will receive the same therapeutic exercise program and sham dry needling.

DETAILED DESCRIPTION:
Therapeutic exercise and dry needling each relieve pain and improve function, but they are different treatment tools.

Therapeutic exercise takes a multitude of forms and results in numerous systemic and local effects, some of which have been investigate among people with knee osteoarthritis. Therapeutic exercise covers a range of targeted physical activities that directly aim to improve muscle strength, neuromotor control, joint range of motion and aerobic fitness. One of the main aims of this therapeutic approach is to improve muscle strength, given that weakness is common in knee osteoarthritis. Enhanced strength of the lower limb may lessen internal knee forces, reduce pain and improve physical function.

Primary knee osteoarthritis provokes pain and disfunction is thought mediated by joint damage and changes in joint homeostasis. Recently, investigations focused in impaired neuromuscular system as a contribution to the above mentioned symptoms in the knee osteoarthritis syndrome explore the use of dry needling. Dry needling is a therapeutic approach for decreasing pain and improve function with high recommended evidence (grade A) effectiveness for upper-quarter myofascial pain, but poorly understood in knee osteoarthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 62 years and older.
* Unilateral or bilateral disfunction and/or knee pain.
* Primary knee ostearthritis fulfilling the American College of Rheumatology criteria for clinical and radiographic diagnostic.
* At least 1 pain point elicited by palpation ipsilateral to the painful knee situated in a taut band of a skeletal muscle of the lower limbs, which usually have referred pain.

Exclusion Criteria:

* Prior diagnoses or prescriptions in the medical record for myopathy or lumbo-sacral neuropathy.
* Previous knee or hip joint replacement surgery of the affected joint.
* Any other surgical procedure of the lower limbs in the previous 6 months.
* Rheumatoid arthritis.
* Initiation of opioid analgesia or cortico-steroid or analgesic injection intervention for hip or knee pain within the previous 30 days.
* Alcohol or drugs consumption.
* Uncontrolled hypertension or moderate to high risk for cardiac complications during exercise.
* Conservative or invasive physical therapy (previous 6 months or during follow-up).
* Taking antiaggregant or anticoagulant medications.
* Physical impairments unrelated to the hip or knee preventing safe participation in exercise, walking or stationary cycling, such as: vision problems that affect mobility, body weight greater than 155 kg, neurogenic disorder, primary or significantly limiting back pain, advanced osteoporosis, or inability to walk 10 metres without an assistive device.
* Inability to comprehend and complete study assessments or comply with study instructions.
* Stated inability to attend or complete the proposed course of intervention and follow-up schedule.
* Fibromyalgia syndrome or other altered affective/cognitive modulation processes of pain perception. .

Ages: 62 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2016-06-16 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Osteoarthritis Index (WOMAC) change assessment. | Base line, through study completion (3 months); and 3, 6 and 12 months follow-up
  The disease-specific questionnaire WOMAC is the most widely used instrument created and validated to evaluate both the symptomatology and function on osteoarthritis of the hip or knee.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Base line, through study completion (3 months); ; and 3, 6 and 12 months follow-up
  Pain intensity will be assessed using a NPRS of 11 points (from 0, no pain, to 10, maximum pain). The patient determined their subjective pain intensity of the painful knee by pointing with 1 of their fingers to mark the level of pain on the scale. .
Barthel Index | Base line, through study completion (3 months); and 3, 6 and 12 months follow-up
  The Barthel Index is considered to be the best of the activities of daily living measurement scales. The modified scoring of the Barthel Index by Shah achieved greater sensitivity and improved reliability than the original version, without causing additional difficulty or affecting the implementation time.
The Timed Up & Go Test | Base line, through study completion (3 months); and 3, 6 and 12 months follow-up
  The patient is asked to perform the rise from a standard arm chair, walk to a line on the floor 3 meters away, turn, return, return and sit down again. The score given is the time taken in seconds to complete the test.
Mini-Mental State Examination (MMSE) | Base line and 12 months follow-up
  It's a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment and to screen for dementia.
EuroQol-5 | Base line, through study completion (3 months); and 3, 6 and 12 months follow-up
  It provides a simple descriptive profile and a single index value for health status through rating of 5 items.

OTHER OUTCOMES:
Total number of falls change assessment. | At Baseline and 1 year follow-up.
  Total number of falls at 1 year follow-up, and to compare with number of falls at one year before the participation on the study.

CONTACTS AND LOCATIONS:
Overall Officials: Eleuterio Atanasio Sánchez Romero, PT, MSc, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez Romero EA, Fernandez-Carnero J, Calvo-Lobo C, Ochoa Saez V, Burgos Caballero V, Pecos-Martin D. Is a Combination of Exercise and Dry Needling Effective for Knee OA? Pain Med. 2020 Feb 1;21(2):349-363. doi: 10.1093/pm/pnz036. PMID 30889250
- See also: website of the University Rey Juan Carlos — http://www.urjc.es